CLINICAL TRIAL: NCT03677362
Title: Weight Loss Intervention in Women With PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 142744
Record Dates: First submitted 2018-09-13; First posted 2018-09-19 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Polycystic Ovary Syndrome; Overweight and Obesity
MeSH Terms: conditions — Polycystic Ovary Syndrome; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Weight loss intervention (Experimental): In the WLI, energy intake will be prescribed at 1200-1500 kcal/d using commercially available portion-controlled entrées, low calorie shakes, fruits/vegetables, and ad-libitum non-caloric beverages. Participants will be asked to consume a minimum daily total of 2 entrées (~200 to 300 kcal each, saturated fat ≤ 3g), 3 shakes (~100 kcal each), five 1-cup servings of fruits/vegetables, and ad libitum non-caloric beverages. Additionally, they will be asked to complete 225 min of moderate intensity PA, and self-monitor diet, PA (self-report) and body weight (home scale) across the 6 mo. intervention. Weekly behavioral counseling sessions (45 min) via Skype will be delivered by a professional health educator (HE) to participants in their homes.
  Interventions: Behavioral: Weight loss intervention

INTERVENTIONS:
Behavioral: Weight loss intervention — In the WLI, energy intake will be prescribed at 1200-1500 kcal/d using commercially available portion-controlled entrées, low calorie shakes, fruits/vegetables, and ad-libitum non-caloric beverages. Participants will be asked to consume a minimum daily total of 2 entrées (~200 to 300 kcal each, saturated fat ≤ 3g), 3 shakes (~100 kcal each), five 1-cup servings of fruits/vegetables, and ad libitum non-caloric beverages. Additionally, they will be asked to complete 225 min of moderate intensity PA, and self-monitor diet, PA (self-report) and body weight (home scale) across the 6 mo. intervention. Weekly behavioral counseling sessions (45 min) via group phone callsSkype will be delivered by a professional health educator (HE) to participants in their homes.

SUMMARY:
The proposed single arm 6 mo. trial will assess the impact of weight loss and fat loss due to a multicomponent remotely-delivered lifestyle intervention on ovulation rates and time-to-ovulation in overweight and obese women with anovulatory infertility caused by PCOS.

DETAILED DESCRIPTION:
Obesity and visceral adiposity are associated with reproductive dysfunction, specifically infertility, problems with ovulation, and decreased rates of conception. Approximately 31% of reproductive aged women in the U.S. are obese. Obese women who become pregnant are at increased risk for miscarriage and pregnancy complications. Infertility treatment using assisted reproductive technologies such as fertility medications, in vitro fertilization or intracytoplasmic sperm injection, is time-intensive, costly, and less effective in obese compared with normal weight women. However, attempts at weight loss to date have been modest at best and the effectiveness of single component hypocaloric diets are questionable. A recently conducted large scale preconception weight loss study in the Netherlands randomized 577 obese infertile women to either a lifestyle intervention prior to fertility treatment or prompt fertility treatment. This study found significantly higher spontaneous pregnancies in the lifestyle intervention group compared to those who promptly received fertility treatment. Additionally, when post hoc analyses were completed on predetermined subgroups, researchers found women with anovulation had more spontaneous pregnancies compared to ovulatory women in the lifestyle intervention group. A few major limitations of this study include: 1) modest weight loss of 4.4 kg and only 38% obtained the minimum goal of 5% weight loss; 2) the study included women with a variety of infertility diagnoses; and 3) limited BMI range of 29-40 kg/m2. More prospective research is necessary to evaluate the effects of weight loss in anovulatory women caused by Polycystic ovarian syndrome (PCOS) as there may be larger benefits in this population such as restoration of ovulation and spontaneous conception. Additionally, there has been limited research investigating fat loss after a lifestyle intervention and the impact on ovulation. Fat loss may play a large role as the purported mechanism by which obesity influences ovulation is through insulin resistance and increased ovarian androgen secretion. Similar to other populations in need of lifestyle interventions, women seeking fertility treatment also have multiple barriers to weight management. Infertility treatment centers in major metropolitan cities often draw individuals from large geographical areas including rural dwelling individuals. Our research team has developed an efficacious weight management program that has shown superior weight loss compared to conventional treatment and has successfully been delivered remotely eliminating concerns of access and transportation and may be well suited for this unique population. However, the acceptability of a remote delivered weight loss intervention, attendance at behavioral sessions, compliance with diet and physical activity (PA) recommendations and self-monitoring (diet, PA, weight), as well as the impact of the magnitude of weight loss on ovulation rates in overweight and obese anovulatory women are unknown, and will be the focus of this study. Over a 2 mo. period, 20 overweight or obese women (BMI > 25 -45 kg/m2, age 21-38 yrs.) seeking initial treatment after 12 mos. of unsuccessful conception (~ 40 new women/mo.) will be recruited to complete a 6 mo. multicomponent weight loss intervention (WLI). Participants must be willing to withhold infertility treatment for the length of the 6 mo. intervention and have the diagnosis of ovulatory dysfunction (anovulation) caused by PCOS as the primary cause of infertility. In the WLI, energy intake will be prescribed at 1200-1500 kcal/d using commercially available portion-controlled entrées, low calorie shakes, fruits/vegetables, and ad-libitum non-caloric beverages. Participants will be asked to consume a minimum daily total of 2 entrées (~200 to 300 kcal each, saturated fat ≤ 3g), 3 shakes (~100 kcal each), five 1-cup servings of fruits/vegetables, and ad libitum non-caloric beverages. Additionally, they will be asked to complete 225 min of moderate intensity PA, and self-monitor diet, PA (self-report) and body weight (home scale) across the 6 mo. intervention. Weekly behavioral counseling sessions (45 min) via Skype will be delivered by a professional health educator (HE) to participants in their homes.

ELIGIBILITY:
Inclusion Criteria:

1. Anovulatory infertility caused by Polycystic ovarian syndrome
2. Age 21 to 42.
3. Body mass index (BMI) > 25 to 45 kg/m2.
4. Weight stable (± 4.6 kg) in previous 3 months
5. Willing to delay fertility treatment for 6 mos

Exclusion Criteria:

1. Unable to participate in moderate-vigorous physical activity (i.e., brisk walking)
2. Currently participating in greater than 3, 30-minute bouts of planned PA/week
3. Participation in a weight loss or PA program in the previous 6 mos.
4. Currently on a weight loss medication (wash out period 2 mos.)
5. Any other infertility diagnosis besides ovulatory dysfunction
6. Binge eating disorder as assessed by the Binge Eating Scale.

Ages: 21 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2020-02-22 (Actual); Study Completion 2020-02-22 (Actual)

PRIMARY OUTCOMES:
Ovulation | 6 months
  Ovulation will be assessed weekly during the 6 mo. intervention by ovulation monitoring kit and the OvuSense device.

SECONDARY OUTCOMES:
Fertility related quality of life | Baseline and 6 months
  The fertility quality of life (FertiQoL) tool (questionnaire)
Body composition | Baseline and 6 months
  A dual energy x-ray absorptiometry scan will determine percent body fat.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Marsh, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gorczyca AM, Steger FL, Ptomey LT, Montgomery RN, Mickelsen R, Smith P, Donnelly JE, Marsh CA. The impact of a group based, remotely delivered weight loss intervention in women with polycystic ovary syndrome on ovulation, quality of life and body composition. Front Reprod Health. 2022 Jul 22;4:940945. doi: 10.3389/frph.2022.940945. eCollection 2022. PMID 36303658